CLINICAL TRIAL: NCT03316495
Title: IMPACT OF PAMPHLET ON THE KNOWLEDGE OF HEALTH EFFECT OF SMOKING: A RANDOMISED CLINICAL TRIAL.
Brief Title: IMPACT OF PAMPHLET ON THE KNOWLEDGE OF HEALTH EFFECT OF SMOKING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Benin (Other)
Collaborators: UBTH (Unknown)
Responsible Party: Principal Investigator, Clement Chinedu Azodo, Head of Department, University of Benin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PAMSMOKE
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- without pamphlet (No Intervention): NOT EXPOSED TO PAMPHLETS
- with pamphlet (Experimental): EXPOSED TO PAMPHLETS
  Interventions: Behavioral: PAMPHLET

INTERVENTIONS:
Behavioral: PAMPHLET — EXPOSURE TO PAMPHLETS
  Arms: with pamphlet

SUMMARY:
Tobacco smoke is one of the most preventable cause of mortality and morbidity worlwide, this study is conducted to compare the knowledge of the health effects of smoking among undergraduates exposed and those not exposed to educational pamphlet. This is designed as a randomized clinical trial among 390 undergraduate in University of Benin Edo State Nigeria. Data collection tool was an interviewer-administered questionnaire. Data obtained would be subjected to regression statistics using IBM SPSS version 21.0. The expected outcome will be a veritable tool in tobacco cessation model.

ELIGIBILITY:
Inclusion Criteria:

- HEALTHY

Exclusion Criteria:

* NOT CONSENTING

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
KNOWLEDGE OF HEALTH EFFECT OF SMOKING | 7 MONTHS
  QUESTIONNAIRE

CONTACTS AND LOCATIONS:
Locations (1):
- Clement Chinedu Azodo, Benin City, Edo, Nigeria